CLINICAL TRIAL: NCT00966069
Title: ReSPeCT: An Unblinded, Randomised, Controlled Trial to Compare Respiratory Sample Collection by a Parent or by a Healthcare Worker at a Home Visit
Brief Title: A Comparison of Respiratory Sample Collection by a Parent or by a Healthcare Worker
Acronym: ReSPeCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Principal Investigator, Dr Stephen Lambert, Senior Research Fellow, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HREC/09/QRCH/42
Record Dates: First submitted 2009-08-24; First posted 2009-08-26 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Tract Infections
Keywords: Respiratory tract infections; Viral infections; Pediatrics; Specimen collection
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthcare worker visit (Active Comparator): Healthcare worker performs home visit when study child has acute respiratory illness to collect a respiratory swab (nasopharyngeal swab).
  At the healthcare worker home visit, the HCW will collect the nasopharyngeal swab, and a parent will collect an anterior nasal swab. The HCW swab is to be returned immediately to the laboratory, and the parent collected swab was placed in a post box for return to the laboratory by surface mail.
  Interventions: Other: Healthcare worker home visit
- Parent collection (Experimental): Home collection of respiratory swab (anterior nose) and mailed return when study subject has an acute respiratory illness.
  Interventions: Other: Parent collection

INTERVENTIONS:
Other: Parent collection — Parent collection of anterior nose specimen when child has an acute respiratory illness, and mailed return of the specimen to the laboratory.
  Arms: Parent collection
Other: Healthcare worker home visit — Healthcare worker performs home visit for collection of respiratory specimen (anterior nose) when study child has an acute respiratory illness.
  Arms: Healthcare worker visit

SUMMARY:
The investigators are aiming to learn more about respiratory infections in young children in the community. To prepare for a larger project, the investigators are conducting this study to get information about the best way to collect and transport respiratory specimens from young children. The investigators would like to test whether parents are more likely to collect a simple respiratory specimen themselves during a child's illness, compared to the likelihood of specimen collection when a home visit is made by a health care worker. Further, the investigators want to compare the likelihood a virus will be identified in both groups.

DETAILED DESCRIPTION:
Prior to this study, there had been one small study conducted in the Netherlands comparing parent-collected specimens at home with collection by a health care worker (HCW) during an arranged home visit. This study suggested that despite there being approximately the same number of illnesses identified in each group, the parent collection group had a higher proportion of ARIs with a specimen collected (43% vs 24%, parent vs HCW home visit), and a higher proportion of specimens tested positive for a virus (80% vs 67%), although neither of these findings was statistically significant.

In order to prepare for a larger, community based study, we would like to test these findings in our environment.

Community-based respiratory infection research has traditionally been conducted by home visit from a health care worker during illness to collect a sample, such as a nasopharyngeal aspirate. This method has the potential to result in non-reporting of illness or failure to collect a specimen due to the invasive nature of specimen collection or the difficulty arranging a home visit time that is convenient for parents and staff. This may bias findings and interfere with generalisability.

Home collection of a simple respiratory sample has recently been demonstrated as an easy and acceptable method of conducting community-based respiratory research. Members of our group were involved in a large, community-based study in Melbourne involving 234 children and their families over a 12-month period. On this study parents successfully kept daily respiratory symptom diaries and collected a combined nose-throat swab when the child had an illness that met the definition for an acute respiratory illness (ARI) of interest. These study methods were acceptable with 87% parents reporting, at the end of the study, they would have been willing to continue with the study for at least another year.

Since that study, parent collection of simple respiratory specimens has been further validated in the hospital setting and used in the home setting.

We have previously shown that a swab combined with viral transport medium-soaked sponge in a secure transport tube is an efficient and safe way of transporting respiratory swabs. The method complies with guidelines for the transport of clinical specimens. As part of this study, we will use this system to allow for the transport of respiratory specimens to the Queensland Paediatric Infectious Diseases (Qpid) Laboratory through the normal surface mail, thereby allowing study families to manage specimen collection and return without the intervention of a study staff member.

Flocked swabs in combination with specific viral transport media have recently been added to specimen collection options, allowing for simple and sensitive specimen collection whilst avoiding more invasive nasopharyngeal aspirates or washes.

With this study, we plan to compare parent and health care worker collection using flocked swabs, and for some specimens they will be returned to the laboratory through normal surface mail.

ELIGIBILITY:
Inclusion Criteria:

* healthy children, 0 to 23 months of age at enrolment (not reached their 2nd birthday)
* born between 36 and 42 weeks gestational age
* written informed consent from parent/guardian (available for telephone contact)
* parent willing to collect an anterior nasal specimen from the study child when meets criteria for ARI of interest

Exclusion Criteria:

* children with chronic pulmonary or cardiovascular disorders (including diagnosed asthma, or frequent use of asthma medication)
* children with chronic metabolic disorders (such as but not limited to diabetes mellitis, renal dysfunction, haemoglobinopathies)
* children with immune system disorders (such as HIV/AIDS or receiving immune system suppressing medications)
* children with other chronic illnesses whose enrolment is deemed by the investigators to make it inappropriate to enrol them onto the study
* parent or guardian with sufficient English language skills to complete study diaries and perform study tasks as required

Max Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of acute respiratory illnesses that have a specimen available for testing in the laboratory. | 6 months
  For this outcome, the Investigators will compare the proportion of all incident ARIs that have a specimen available for testing in each group (HCW vs parent collection).

SECONDARY OUTCOMES:
Proportion of specimens collected that have a virus able to be detected. | 6 months
  For this outcome, the Investigators will compare the proportion of all specimens collected during incident ARIs in each group (HCW vs parent collection) that have any virus detected.
Proportion of swabs collected at home visit with virus detected (HCW nasopharyngeal swab vs parent collected anterior nose swab). | 6 months
  This comparison is restricted to children randomised to the health care worker collection group. In this group, at the home visit the HCW will collect a nasopharyngeal swab, place it in universal transport media, and return it immediately to the laboratory. At the same home visit, a parent will collect a dry anterior nasal swab, it will be placed in a post box near the subject's home, and returned to the laboratory by normal surface mail. For this outcome, the Investigators will compare the proportion of all specimens collected during incident ARIs in the HCW group that have any virus detected (HCW nasopharyngeal swab vs parent collected anterior nose swab).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Grimwood, MD, Principal Investigator — The University of Queensland; Theo P Sloots, PhD, Principal Investigator — Queensland Paediatric Infectious Diseases Laboratory; Michael D Nissen, FRACP, Principal Investigator — Queensland Paediatric Infectious Disease Laboratory; Stephen B Lambert, MBBS, Principal Investigator — Queensland Paediatric Infectious Diseases Laboratory
Locations (1):
- Queensland Children's Medical Research Institute, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zoch-Lesniak B, Ware RS, Grimwood K, Lambert SB. The Respiratory Specimen Collection Trial (ReSpeCT): A Randomized Controlled Trial to Compare Quality and Timeliness of Respiratory Sample Collection in the Home by Parents and Healthcare Workers From Children Aged <2 Years. J Pediatric Infect Dis Soc. 2020 Apr 30;9(2):134-141. doi: 10.1093/jpids/piy136. PMID 30657971